CLINICAL TRIAL: NCT05125081
Title: RCT Study of Liuwei Dihuang Pill Preventing and Treating Presbycusis With Shen (Kidney)-Yin Deficiency
Brief Title: Efficacy and Safety of Liuwei Dihuang Pill Versus Placebo in Presbycusis With Shen (Kidney)-Yin Deficiency
Acronym: RLDP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jianrong Shi, Professor&Vice-Principal, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLDP-2021
Record Dates: First submitted 2021-11-17; First posted 2021-11-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Presbycusis; Age-related Hearing Loss; Hearing Disorders and Deafness
Keywords: Presbycusis; Age-related hearing loss; Liuwei Dihuang Pill
MeSH Terms: conditions — Presbycusis; Hearing Disorders; Deafness | interventions — Liuwei Dihuang Decoction

STUDY DESIGN:
Intervention Model Description: A Phase 2 Randomized, Double-blind, Placebo-controlled, Multicenter Study of Liuwei Dihuang Pill Administered by taking orally in Adults With Presbycusis With Shen (Kidney)-Yin Deficiency.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDP group (Experimental): Liuwei Dihuang Pill (LDP）marketed product in China donated by pharmaceutical company.
  Interventions: Drug: Liuwei Dihuang Pill (marketed product in China)
- placebo group (Placebo Comparator): Same smell, color and shape as Liuwei Dihuang Pill (LDP）without herbs in capsules.
  Interventions: Drug: Liuwei Dihuang Pill（placebo ）

INTERVENTIONS:
Drug: Liuwei Dihuang Pill (marketed product in China) — LDP group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo group and LDP group. The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the LDP group and placebo group at a ratio of 1:1. The drug was administered for 48 weeks, 3 times a day, 8 pills each time.
  Other Names: Liu Wei Di Huang Pill
  Arms: LDP group
Drug: Liuwei Dihuang Pill（placebo ） — LDP group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo group and LDP group. The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the LDP group and placebo group at a ratio of 1:1. The drug was administered for 48 weeks, 3 times a day, 8 pills each time.
  Other Names: placebo group
  Arms: placebo group

SUMMARY:
The objective of this study is to examine the effects and safety of Liuwei Dihuang pill and placebo in presbycusis with Shen (kidney)-yin deficiency.

DETAILED DESCRIPTION:
There are no approved pharmacologic therapies for age-related hearing loss (ARHL), also known as presbycusis. Based on the syndrome differentiation in Chinese medicine (CM) theory, the pathogenesis of presbycusis is related to the Shen (kidney)-yin deficiency. Liuwei Dihuang Pill (LDP) is effective and commonly prescribed for the treatment of Shen-yin deficiency.

The main purpose of this study is to try to demonstrate an improvement in phonetically balanced maximum (PBmax) after 1 years of treatment with the LDP versus the placebo. Subjects will undergo a safety follow-up after the treatment period. Safety and efficacy will be determined by looking at a number of assessments (physical examinations, blood sampling, hearing assessments, questionnaires, etc.).The amount of drug in the blood will also be measured.

It is expected that around 120 people (at least 60 in each arm) with presbycusis with Shen (kidney)-yin deficiency may take part in the study. The study participants will be recruited at around 6 sites in the Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a current diagnosis of presbyacusis with symmetrical hearing loss, defined as 15-dB or less difference in pure tone average between ears at 0.5, 1, 2 and 4kHz. The average hearing threshold loss level is mild or moderate (20 ≤ average hearing threshold < 50 dBHL).
2. Adult aged 65-75 years inclusive.
3. Maximum speech recognition rate in quiet environment is equal to or over 60% with ability to communicate well.
4. Subjects have no cognitive impairment with CDR score =0.
5. Subjects must have a current diagnosis of Shen (Kidney)-Yin Deficiency.
6. Subjects have read and voluntarily signed the Informed Consent Form (ICF) after all questions have been answered and prior to any study-mandated procedure.

Exclusion Criteria:

1. Subjects with sudden hearing loss or pure tone hearing fluctuation within the three months.
2. Subjects with a history of serious mental illness.
3. Subjects with severe cardiac insufficiency, malignant tumor or other serious systemic diseases.
4. Subjects with conductive deafness, congenital deafness, hereditary deafness, inner ear immune and autoimmune inner ear diseases, auditory neuropathy, toxic deafness and noise deafness.
5. Subjects with organic ear diseases, abnormal ear structure and symptomatic cerebral infarction.
6. Subjects with dementia, neurosyphilis, hypothyroidism and depression.
7. Subjects has previously participated in other clinical trial within the three months.
8. Subjects with using hearing aids or devices.
9. Other situations where the researcher thinks it is inappropriate to participate in this research.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Change in PB-Max after 48 weeks of treatment | 48 weeks
  To compare the change in PB-Max using the Word Recognition in Quiet test measured with Consonant-Nucleus-Consonant (CNC) word lists from baseline (week 1 to week 48) between LDP and placebo.

SECONDARY OUTCOMES:
Change in Speech recognition threshold (SRT) after 24 weeks and 48 weeks of treatment | 24 weeks，48 weeks
  To compare the change in Speech recognition threshold (SRT) using the Word Recognition in Quiet test measured with Consonant-Nucleus-Consonant (CNC) word lists from baseline (week 1 to week 24，week 48) between LDP and placebo.
Change in Pure Tone Average (PTA) after 24 weeks and 48 weeks of treatment | 24 weeks，48 weeks
  To compare the change in Pure Tone Average (PTA) using the Air conduction audiometry for hearing at certain range (Hz) from baseline (week 1 to week 24，week 48) between LDP and placebo.
Change in Shen (Kidney)-Yin Deficiency Syndrome Questionnaire after 12 weeks，24 weeks，36 weeks and 48 weeks of treatment | 12 weeks，24 weeks，36 weeks，48 weeks
  To compare the change in Shen (Kidney)-Yin Deficiency Syndrome Questionnaire using Face to face Interview for the scores from baseline (week 1 to week 12，week 24，week 36 and week 48) between LDP and placebo (range, 0 [best] to 100 [worst]).
Change in Tinnitus Handicap Inventory（THI）after 12 weeks，24 weeks，36 weeks and 48 weeks of treatment | 12 weeks，24 weeks，36 weeks，48 weeks
  To compare the change in Tinnitus Handicap Inventory（THI）using Face to face Interview for the scores from baseline (week 1 to week 12，week 24，week 36 and week 48) between LDP and placebo (range, 0 [best] to 100 [worst]).
Change in Mini-mental State Examination (MMSE) after 12 weeks，24 weeks，36 weeks and 48 weeks of treatment | 12 weeks，24 weeks，36 weeks，48 weeks
  To compare the change in Mini-mental State Examination (MMSE) using Face to face Interview for the scores from baseline (week 1 to week 12，week 24，week 36 and week 48) between LDP and placebo (range, 0 [worst] to 100 [best]).

OTHER OUTCOMES:
Change in ABR after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of auditory brainstem response（ABR ）from baseline (week 1 to week 48) between LDP and placebo.
Change in DPOAE pass rate after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the pass rate levels of distortion product otoacoustic emissions（DPOAE）from baseline (week 1 to week 48) between LDP and placebo.
Change in serum CRP after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum C-reactive protein (CRP) related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum cytokines after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum cytokines related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in Peripheral Blood Mononuclear Cells after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of Peripheral Blood Mononuclear Cells related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum MDA after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum Malondialdehyde (MDA) related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum MPO after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum Myeloperoxidase (MPO) related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum GSH after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum L-Glutathione(GSH) related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum T-AOC after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum Total antioxidant capacity（T-AOC）related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in serum NfL after 48 weeks of treatment | 48 weeks
  The absolute values of changes in the levels of serum Neurofilament Light（NfL）related to the mechanism from baseline (week 1 to week 48) between LDP and placebo.
Change in Composite indictors after 48 weeks of treatment | 48 weeks
  To compare the changes in Composite indictors (some individual indicators are compiled into a single index on the basis of an underlying model according to specific evaluation) from baseline (week 1 to week 48) between LDP and placebo.
Change in hemodynamic signals of resting fMRI after 48 weeks of treatment | 48 weeks
  The changes in hemodynamic signals of resting functional magnetic resonance imaging (fMRI) related to the mechanism from baseline (week 1 to week 48) between LDP and placebo. 40 patients were selected for this study.
Change in perpheral metabolomics after 48 weeks of treatment | 48 weeks
  To compare the change in perpheral metabolomics from baseline(week 1 to week 48) between LDP and placebo.
Change in perpheral proteomics after 48 weeks of treatment | 48 weeks
  To compare the change in perpheral proteomics from baseline(week 1 to week 48) between LDP and placebo.
Adverse Events | 24 weeks，48 weeks
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jianrong Shi, Doctor, Study Director — Shanghai Jiao Tong University School of Medicine; Jianning Zhang, Doctor, Principal Investigator — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine; Ping Huang, Doctor, Principal Investigator — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine; Hongsheng Tan, Doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (6):
- China (6):
  - Community Health Service Center of North Sichuan Road, Hongkou District, Shanghai, Shanghai, Shanghai Municipality
  - Jiaxing Street Community Health Service Center, Hongkou District, Shanghai, Shanghai, Shanghai Municipality
  - Community Health Service Center of Tianlin Street, Xuhui District, Shanghai, Shanghai, Shanghai Municipality
  - Sixth people's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Juquan New Town Community Health Service Center, Gucun Town, Baoshan District, Shanghai, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Bednar MM, DeMartinis N, Banerjee A, Bowditch S, Gaudreault F, Zumpano L, Lin FR. The Safety and Efficacy of PF-04958242 in Age-Related Sensorineural Hearing Loss: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Jul;141(7):607-13. doi: 10.1001/jamaoto.2015.0791. PMID 25997115
- [Background] McLean WJ, Hinton AS, Herby JTJ, Salt AN, Hartsock JJ, Wilson S, Lucchino DL, Lenarz T, Warnecke A, Prenzler N, Schmitt H, King S, Jackson LE, Rosenbloom J, Atiee G, Bear M, Runge CL, Gifford RH, Rauch SD, Lee DJ, Langer R, Karp JM, Loose C, LeBel C. Improved Speech Intelligibility in Subjects With Stable Sensorineural Hearing Loss Following Intratympanic Dosing of FX-322 in a Phase 1b Study. Otol Neurotol. 2021 Aug 1;42(7):e849-e857. doi: 10.1097/MAO.0000000000003120. PMID 33617194
- [Background] Ge JR, Xie LH, Chen J, Li SQ, Xu HJ, Lai YL, Qiu LL, Ni CB. Liuwei Dihuang Pill () Treats Postmenopausal Osteoporosis with Shen (Kidney) Yin Deficiency via Janus Kinase/Signal Transducer and Activator of Transcription Signal Pathway by Up-regulating Cardiotrophin-Like Cytokine Factor 1 Expression. Chin J Integr Med. 2018 Jun;24(6):415-422. doi: 10.1007/s11655-016-2744-2. Epub 2016 Dec 27. PMID 28028720
- See also: 《The World Report on Hearing》2021 — https://www.who.int/publications/i/item/world-report-on-hearing